CLINICAL TRIAL: NCT05204979
Title: Vaginal Versus Sublingual Misoprostol Before Intrauterine Device Insertion in Women With Pervious Caesarian Section
Brief Title: Vaginal Vs Subling Misoprost Before Iud Insertion in Women With Previous CS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rofida Mohamed Arafa Taha, Director, Ain Shams University
Other Study IDs: THESIS FOR PARTIA
Record Dates: First submitted 2021-06-23; First posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: IUD Insertion
Keywords: Misoprostol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Misopristol: Group A: vaginal misoprostol will be taken Group B: sublingual misoprostol will be taken
  Interventions: Other: Vaginal Versus Sublingual misoprostol

INTERVENTIONS:
Other: Vaginal Versus Sublingual misoprostol — Insertion failures of intra uterine devices and cervical problems seem to occur more often among women who have never delivered vaginally. Several studies have shown the benefit of misoprostol as a cervical ripening agent in nonpregnant women. This trial will compare the effect of vaginal versus sublingual misoprostol prior to insertion of an intrauterine device in multiparous women delivered by CS.

SUMMARY:
Insertion failures of intrauterine devices and cervical problems seem to occur more often among women who have never delivered vaginally. This trial will compare the effect of vaginal versus sublingual misoprostol prior to insertion of an intrauterine device in multiparous women delivered by CS.

DETAILED DESCRIPTION:
Intrauterine devices (IUDs) are widely used as reversible contraceptives. The current use of IUDs among reproductive-aged women ranges from 8 to 15% worldwide. Reported complications related to IUD insertion are 8.8% insertion failure, 2.8-11.5% cervical problems, 0.2% cervical perforation, 0.2% syncope and 5.8% expulsion. Insertion failures and cervical problems seem to occur more often among women who have never delivered vaginally.

Misoprostol is an inexpensive PGE1. Priming with misoprostol prior to hysteroscopy and dilatation and curettage (D&C) in premenopausal women resulted in an increased cervical dilatation and rate of cervical laceration. Moreover, several studies have shown the benefit of misoprostol as a cervical ripening agent in nonpregnant women. The effect of misoprostol is dependent on the route of administration. Sublingual administration of misoprostol has been shown to be more effective also for cervical priming compared with oral administration and equally effective as vaginal administration.

larger studies on the effect of misoprostol for IUD insertion are lacking. Investigator therefore will conduct a trial aiming to compare the effect of vaginal versus sublingual misoprostol prior to insertion of an intrauterine device in multiparous women delivered by CS.

ELIGIBILITY:
Inclusion Criteria:

Women at the reproductive age group between 20-40 years Women who previously delivered by cesarean section. Women with BMI between 20- 30.

Exclusion Criteria:

Women had a previous vaginal operations. Women with contraindications for misoprostol use (pregnancy, prostaglandin allergy) Women with a contraindication for IUCD insertion (e.g., less than sex weeks post-partum, gynecologic malignancy, uterine bleeding of undetermined origin, fibroids or other uterine abnormalities, active vaginitis or cervicitis, a history of PID or puerperal sepsis).

Women on anticoagulant therapy or having any coagulopathy. Women who refused to participate.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women
Study Population: The study will be conducted on multiparous women delivered only by CS seeking intra uterine device insertion
Sampling Method: Probability Sample
Enrollment: 2 (Estimated)
Dates: Start 2021-06-23 (Actual); Primary Completion 2022-02-17 (Estimated); Study Completion 2022-05-25 (Estimated)

PRIMARY OUTCOMES:
The proportion of easy IUD Insertion | 24 hours
  Difficulty of IUD insertion will be measured by cervical dilatation that determined by two factors:
  1. Degree of dilatation of cervix by using gradual Hegar 1, 2, 3.
  2. The degree of difficulty of the IUD insertion judged as the resistance of the internal cervical os experienced by the investigator and classified as 'easy', 'moderate' or 'difficult'.
  [Time Frame: Easy: Using Hegar 3 and easy of difficulty of insertion. Moderate: Using Hegar 2 and moderate of difficulty of insertion. Difficult: Using Hegar 1 and difficult of difficulty of insertion]

SECONDARY OUTCOMES:
the pain during insertion | 24 hours
  Pain will be measured using a visual analog scale (VAS) pain score reported by participants during IUD insertion. Pain score will be measured using a visual analogue scale consisting of a 10 cm horizontal straight line on which 0 cm corresponds to no pain and 10 cm to the worst pain. VAS is rated as 0 no pain. 1-3 for mild pain. 4-6 for average pain and 7-9 for severe pain and 10 for extremely sever pain an individual can experience.

CONTACTS AND LOCATIONS:
Overall Officials: Hassan MD awad, consultant, Study Chair — professor; Rofida M Taha, doctor, Study Chair — doctor
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No